CLINICAL TRIAL: NCT01409226
Title: A Study to Evaluate 3.0 Tesla Magnetic Resonance Imaging of the Breasts in High Risk Women
Brief Title: 3.0 Tesla Magnetic Resonance Imaging for Breast Cancer Detection in High Risk Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-0051
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: high-risk of breast cancer; BRCA1 mutation carrier; BRCA2 mutation carrier; diagnostic; MRI; BI-RADS 4; mammographically occult
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Biopsy

ARMS (1):
- MRI (Experimental)
  Interventions: Device: 3.0-T MRI; Procedure: biopsy

INTERVENTIONS:
Device: 3.0-T MRI — Participants undergo MRI prior to biopsy.
Procedure: biopsy — Participants undergo breast biopsy after 3.0-T MRI.

SUMMARY:
This study is to find out if 3.0 Tesla (3.0-T) Magnetic Resonance Imaging (MRI) will improve in diagnosing breast cancer in women with high-risk of breast cancer.

DETAILED DESCRIPTION:
Life time risk of developing breast cancer is greatly elevated in women with familial breast cancer, especially in BRCA carriers. Prevention and early detection strategies in these high risk women include risk reducing surgery, chemoprevention and close surveillance with semiannual clinical breast exams and yearly mammograms starting at age 25-35. Unfortunately, screening mammography detects only half the breast cancers in mutation carriers, presumably due to higher breast density in the younger women and perhaps due to inherent characteristics of their tumors such as rapid growth. In light of these limitations in this high risk group, some have suggested incorporation of semiannual mammograms and/or other imaging modalities such as ultrasound (US) and MRI.

In this study, high risk women who have a suspicious mammographic lesion - categorized as Breast Imaging Reporting and data System (BI-RADS) 4 will be recruited to undergo a breast MRI before to a biopsy of the suspicious abnormality. All women will undergo a biopsy as a part of her standard of care. The results of the MRI will not influence our decision on whether a biopsy should be performed. The MRI results will be compared with the biopsy results with pathology as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Women at high risk of developing breast cancer as outlined by the American Cancer society (ACS): women with known predisposing mutations (in BRCA1, 2 or PTEN genes), women with first degree relative who is a known carrier or has a 20% or more life time risk of breast cancer.
* The above high-risk women with a suspicious lesion classified as BIRADS 4 that is detected on mammography. Since the spatial resolution of 3.0-T breast MRI is similar to digital mammography, there is no limitation to the size of the mammographic lesion.

Exclusion Criteria:

* Pregnancy or lactating women
* Contraindications for MRI:

  1. electrical implants (e.g. cardiac pacemakers or perfusion pumps)
  2. ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  3. pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
  4. weight over 350 lbs
* Although a women meets our criteria for high risks for breast cancer and has an abnormal mammogram, she will be excluded from our study if her insurer does not provide payment for the breast MRI. The suspicious lesion will be biopsied under mammographic guidance as part of her standard of care. The third party carriers have been reimbursing payment for a breast MRI in these high risk women, especially after the ACS guidelines were released in 2007. Therefore, this outcome is unlikely to occur.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with mammographically occult breast cancer detected by 3.0-T MRI | 2 years
  This is the frequency of mammographically occult breast cancer detected by 3.0-T MRI in a subset of high risk women with a suspicious mammographically detected lesion.

SECONDARY OUTCOMES:
Percentage of participants with incidental lesions detected by MRI | 2 years
  This is defined as the number of participants who have incidental lesions by MRI over the total number of participants.
  Incidental lesions are the lesions only detected by 3.0-T MRI, and not seen by mammography.
False positive rate | 2 years
  The rate is defined as the percentage of participants who are diagnosed with breast cancer by MRI, yet not have the cancer. The MRI results will be compared with biopsy results with the pathology as the gold standard.
False negative rate | 2 years
  The rate is defined as the percentage of participants who are diagnosed by pathology, yet not by MRI. The MRI results will be compared with biopsy results with the pathology as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Moy, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Medical Center, New York, New York, United States